CLINICAL TRIAL: NCT03128229
Title: Diabetic Kidney Alarm (DKA) Study - Tubulopathy in Diabetic Ketoacidosis
Brief Title: Diabetic Kidney Alarm (DKA) Study
Acronym: DKA
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1403
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes Mellitus; Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine collection at 0-8h and 12-24h after starting IV insulin, and at 3 month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overarching goals of this study are to determine whether tubular dysfunction (elevated urine sodium, bicarbonate and amino acids) and injury (elevated kidney injury molecule 1 [KIM-1], neutrophil gelatinase-associated lipocalin [NGAL] and matrix metallopeptidase 9 [MMP9]) exist in diabetic ketoacidosis (age 3-18), whether it is reversible and whether it is related to uricosuria and copeptin. The investigators propose to study a cohort of youth (ages 3-18, n=40) with T1D who have serum and urine collection at DKA diagnosis and 3-month follow-up.

DETAILED DESCRIPTION:
Every year over 86,000 children (0-14 years) worldwide are diagnosed with type 1 diabetes (T1D) translating to a lifetime of exposure and risk for early death from cardiovascular disease (CVD) and diabetic kidney disease (DKD). DKD, which manifests in children and adolescents, remains the leading cause of renal failure and dialysis in the Western world (4). While diabetic glomerulopathy has received significant attention from researchers, determinants of tubular injury in diabetes are less well examined. Compared to glomerular injury, tubular injury is known to associate better with renal function. The majority of youth diagnosed with T1D in the US present with diabetic ketoacidosis (DKA), a condition associated with risks factors for tubular injury including dehydration, metabolic acidosis and acute glycemia. It is unknown whether DKA is associated with tubular injury. The investigators published the first report showing that youth with established T1D have more acidic urine and higher fractional excretion of uric acid (FeUA) than their non-diabetic peers, which may predispose to UUA-mediated tubulopathy. Furthermore, T1D is associated with vasopressin overactivity, and the investigators reported strong relationships between serum copeptin, a reliable surrogate marker for vasopressin, and DKD in T1D. The overarching goals of this study are to determine whether tubular dysfunction (elevated urine sodium, bicarbonate and amino acids) and injury (elevated KIM-1, NGAL and MMP9) exist in DKA, whether it is reversible and whether it is related to uricosuria and copeptin. The investigators propose to study a cohort of youth (ages 3-18, n=40) with T1D who have serum and urine collection at DKA diagnosis and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* New onset T1D and known T1D
* DKA (mild, moderate and severe DKA eligible)
* 3-17 years of age
* Toilet trained
* Boys and girls
* All ethnicities
* Initial presentation to Children's Hospital Colorado (CHCO) Main ED

Exclusion Criteria:

* Non-T1D etiology
* History of chronic kidney disease (eGFR <60ml/min/1.73m2) or dialysis dependent
* History of tubulopathy (e.g. Fanconi syndrome)
* Currently menstruating
* Patient visiting Colorado with plan to establish diabetes care outside of Colorado
* On ACE-inhibitors or angiotensin II-receptor blockers (ARB)
* On sodium-glucose co-transporter 2 inhibitors (SGLT2 inhibitors)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants (3-18 years) with T1D presenting with DKA will be recruited from the Emergency Department (ED) at Children's Hospital Colorado.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Proximal tubular dysfunction | At DKA (0-8 and 12-24 hours after starting IV insulin)
  Change in urine Na, HCO3 and amino acids concentrations
Proximal tubular injury | At DKA (0-8 and 12-24 hours after starting IV insulin)
  Change in urine and serum NGAL, KIM-1 and MMP9 concentrations

SECONDARY OUTCOMES:
Proposed mediators of tubular dysfunction and injury | At DKA (0-8 and 12-24 hours after starting IV insulin)
  Change in urine uric acid and serum fructose.
Proposed mediators of tubular dysfunction and injury | At DKA (0-8 hours after starting IV insulin)
  Presence of urine uric acid crystals by polarized microscopy
Proposed mediators of tubular dysfunction and injury | At DKA (12-24 hours after starting IV insulin)
  Presence of urine uric acid crystals by polarized microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjornstad P, Johnson RJ, Snell-Bergeon JK, Pyle L, Davis A, Foster N, Cherney DZ, Maahs DM. Albuminuria is associated with greater copeptin concentrations in men with type 1 diabetes: A brief report from the T1D exchange Biobank. J Diabetes Complications. 2017 Feb;31(2):387-389. doi: 10.1016/j.jdiacomp.2016.11.015. Epub 2016 Dec 7. PMID 27979439
- [Background] Bjornstad P, Maahs DM, Jensen T, Lanaspa MA, Johnson RJ, Rewers M, Snell-Bergeon JK. Elevated copeptin is associated with atherosclerosis and diabetic kidney disease in adults with type 1 diabetes. J Diabetes Complications. 2016 Aug;30(6):1093-6. doi: 10.1016/j.jdiacomp.2016.04.012. Epub 2016 Apr 19. PMID 27141815
- [Background] Roncal-Jimenez CA, Milagres T, Andres-Hernando A, Kuwabara M, Jensen T, Song Z, Bjornstad P, Garcia GE, Sato Y, Sanchez-Lozada LG, Lanaspa MA, Johnson RJ. Effects of exogenous desmopressin on a model of heat stress nephropathy in mice. Am J Physiol Renal Physiol. 2017 Mar 1;312(3):F418-F426. doi: 10.1152/ajprenal.00495.2016. Epub 2016 Dec 21. PMID 28003190
- [Background] Bakes K, Haukoos JS, Deakyne SJ, Hopkins E, Easter J, McFann K, Brent A, Rewers A. Effect of Volume of Fluid Resuscitation on Metabolic Normalization in Children Presenting in Diabetic Ketoacidosis: A Randomized Controlled Trial. J Emerg Med. 2016 Apr;50(4):551-9. doi: 10.1016/j.jemermed.2015.12.003. Epub 2016 Jan 25. PMID 26823137
- [Background] Rewers A, Dong F, Slover RH, Klingensmith GJ, Rewers M. Incidence of diabetic ketoacidosis at diagnosis of type 1 diabetes in Colorado youth, 1998-2012. JAMA. 2015 Apr 21;313(15):1570-2. doi: 10.1001/jama.2015.1414. No abstract available. PMID 25898057
- [Background] Dabelea D, Rewers A, Stafford JM, Standiford DA, Lawrence JM, Saydah S, Imperatore G, D'Agostino RB Jr, Mayer-Davis EJ, Pihoker C; SEARCH for Diabetes in Youth Study Group. Trends in the prevalence of ketoacidosis at diabetes diagnosis: the SEARCH for diabetes in youth study. Pediatrics. 2014 Apr;133(4):e938-45. doi: 10.1542/peds.2013-2795. Epub 2014 Mar 31. PMID 24685959
- [Background] Rewers A, Chase HP, Mackenzie T, Walravens P, Roback M, Rewers M, Hamman RF, Klingensmith G. Predictors of acute complications in children with type 1 diabetes. JAMA. 2002 May 15;287(19):2511-8. doi: 10.1001/jama.287.19.2511. PMID 12020331
- [Background] Bjornstad P, Roncal C, Milagres T, Pyle L, Lanaspa MA, Bishop FK, Snell-Bergeon JK, Johnson RJ, Wadwa RP, Maahs DM. Hyperfiltration and uricosuria in adolescents with type 1 diabetes. Pediatr Nephrol. 2016 May;31(5):787-93. doi: 10.1007/s00467-015-3299-8. Epub 2015 Dec 23. PMID 26701836